CLINICAL TRIAL: NCT03530605
Title: Use of Optune TTF With Radiation as an Alternative for Elderly Patients With Primary CNS Lymphoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never initiated, PI left institution
Sponsor: Saint Luke's Health System (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Optune TTF in PCNSL
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Central Nervous System Neoplasms, Primary
Keywords: PCNSL, primary central nervous system lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Intervention Model Description: prospective group (non-randomized) compared to historical matched controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Optune TTF Device (Experimental): Optune TTF treatment
  Interventions: Device: Optune TTF device
- Historical matched control (No Intervention): age-matched historical controls

INTERVENTIONS:
Device: Optune TTF device — portable device which produces electrical fields
  Arms: Optune TTF Device

SUMMARY:
This study will compare the overall survival (OS) time of elderly patients who would not tolerate standard chemotherapy for PCNSL treated with WBXRT together with Optune-TTF to those treated with whole-brain radiotherapy alone.

Standard treatment of primary central nervous system lymphoma (PCNSL) for patients with good performance status involves high-dose methotrexate-based chemotherapy regimens and whole-brain radiation therapy (WBXRT). Although up to 20% of patients with PCNSL are 80 years of age or older, little data exist with regard to optimal treatment of this patient population and they often do not qualify for clinical trials. In addition, elderly patients have a poorer rate of complete and partial response and increased risk of toxicity when treated with standard chemotherapy regimens. Though a consensus does not exist, radiotherapy alone is often used in these patients to minimize toxic effects of more aggressive chemotherapies.

The Optune TTF device has proven effective in treating high-grade gliomas and is currently being investigated to treat meningiomas and metastatic lesions in the brain as well as other tumor types elsewhere in the body. It is generally well tolerated with no known systemic side effects, producing only an occasional local skin reaction. The mechanism of action is independent of tumor type and therefore may be effective in treating lymphoma as well.

ELIGIBILITY:
Inclusion Criteria:

* Histological de novo diagnosis of PCNSL
* Tumor located in the supra-tentorial brain region
* Karnofsky performance score of 70 or above
* Ineligible for chemotherapy due to age or other co-morbidities
* Life expectancy of at least 3 months
* Patient has a caretaker willing to assist with study compliance
* Patient is able to provide written consent on their own behalf

Exclusion Criteria:

* Second or subsequent recurrence of PCNSL
* Patient wishes to receive systemic treatment
* Implanted electronic medical device in the brain (deep brain stimulator, vagus nerve stimulator, programmable shunt, etc.)
* Skull defect without replacement
* Prior radiation, surgery, or chemotherapy for PCNSL within the 4 weeks prior to enrollment
* Patient unable to comply with Optune device treatment or the study follow- up schedule
* Active participation in another therapeutic clinical trial
* Patient unable to provide written consent on their own behalf

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival Time | 4 years
  Overall survival time

SECONDARY OUTCOMES:
Progression-Free Survival Time | 2 years
  Progression-free survival time
One-Year Survival Rate | 1 year
  One-year survival rate
Radiographic Response Rate | 2 years
  Tumor response by MRI measurement
Steroid & Antiepileptic Use | 2 years
  use of concomitant steroids and antiepileptic use